CLINICAL TRIAL: NCT06819982
Title: Autonome À Domicile Grâce À Un Appareil Connecté Et À Un Suivi Ergo
Brief Title: Autonomous At Home with Occupational Therapy Support and Assistive Devices
Acronym: AUDACE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: AUDACE
Record Dates: First submitted 2025-01-28; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-01

CONDITIONS: Frailty; Aging; Home Care Services
Keywords: Education, Continuing; Home Care Services; Monitoring, Ambulatory; Occupational Therapy; Personal Autonomy; Primary Health Care / methods; Program Evaluation; Self-Help Devices
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BCM2.0 (Experimental): The BCM2.0 programme provides occupational therapy sessions and assistive devices to support older people who want to age in place.
  Interventions: Other: BCM2.0

INTERVENTIONS:
Other: BCM2.0 — The BCM2.0 programme provides occupational therapy sessions and assistive devices to support older people who want to age in place.

SUMMARY:
The aim of the AUDACE study is to evaluate the 'Bien chez Moi 2.0' programme, to assess how, for whom and why do assistive devices, integrated with occupational therapy support, enable older people to remain at home, and under what conditions? The study assesses the impact on areas such as the degree of autonomy, the extent to which life goals are taken into account, the feeling of security at home, the use of hospital emergency services and the postponement of definitive institutionalisation in a nursing home. The expected results of this study are to be able to robustly describe the impact of the 'Bien chez moi 2.0' programme in the areas listed above.

DETAILED DESCRIPTION:
Background The BCM2.0 programme provides occupational therapy sessions and assistive devices to support older people who want to age in place. The investigators designed the AUDACE evaluation to improve understanding of the programme and its effectiveness, and to promote a favourable context for the professional empowerment of occupational therapists as primary care providers.

Methods The investigators involved home care occupational therapists at every stage of the protocol design to ensure that the tools, training, and organisational structures put in place for the evaluation could also form the basis of their routine practice, harmonising their practices, ethos and processes.

The investigators designed a realist mixed methods evaluation to answer the following question: "How, for whom and why do assistive devices, integrated with occupational therapy support, enable older people to remain at home, and under what conditions?" Interrelated components addressed different research sub-questions: (1a) To describe the evaluation population, interventions, and contexts: a descriptive quantitative study using baseline data from all BCM2.0 beneficiaries. (1b) To describe the frailty process in older people receiving the programme: a qualitative study using semi-structured individual interviews with a biographical dimension. (2) To explore the enrolment process: focus groups with occupational therapists, following a realist approach. (3) To assess effectiveness: a prospective cohort study with up to 12 months follow-up of all BCM2.0 beneficiaries. (4) To identify barriers and facilitators to implementation: multiple nested case study in five areas, using a realist approach. (5) To build a learning community to clarify ethical considerations: communities of practice meetings.

ELIGIBILITY:
Inclusion Criteria:

* people aged 65 and over
* living at home in the Walloon and Brussels regions
* who are considered frail or at risk of frailty. The risk of frailty is defined as having at least one loss of intrinsic capacity measured by a trained occupational therapist using the ICOPE screening tool

Exclusion Criteria:

* People benefiting from other AViQ autonomy programmes of this project are excluded

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 3900 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2025-09-04 (Estimated); Study Completion 2025-09-04 (Estimated)

PRIMARY OUTCOMES:
COPM | At enrolment and six months follow up.
  Endpoints will be calculated as the within-subject difference in measurement between baseline and six-month follow-up in Canadian Occupational Performance Measure (COPM), assessing daily occupations of importance that people are unable to perform.
  Scale description:
  Canadian Occupational Performance Measure Range 1-10 Higher score = Better outcome

SECONDARY OUTCOMES:
Short FES-I | At enrolment and six months follow up.
  Endpoint will be calculated as the within-subject difference in measurement between baseline and six-month follow-up for short FES-I (short Fall efficacy scale - international, measuring concern over the possibility of falling)
  Scale description:
  short Fall efficacy scale - international Range 7-28 Higher score = Worse outcome
Health-related QoL | At enrolment and six months follow up.
  Endpoint will be calculated as the within-subject difference in measurement between baseline and six-month follow-up for EQ-5D-5L mapped to Belgian utility scores.
  Scale description:
  EQ-5D-5L Range: Below 0 to 1 Higher score = Better outcome
Hospitalisation | At enrolment and six months follow up.
  Endpoint will be calculated as the within-subject difference in measurement between baseline and six-month follow-up for use of hospitalisation and institutionalisation in a nursing home (number of stay in the last six months).
  Scale description:
  Number of stay in hospital or nursing home Range: 0+ Higher score = Worse outcome
Use of assistive devices | At enrolment and six months follow up.
  Endpoint will be calculated as the within-subject difference in measurement between baseline and six-month follow-up for use of assistive devices (binary response).
Sense of security | At enrolment and six months follow up.
  Endpoint will be calculated as the within-subject difference in measurement between baseline and six-month follow-up for sense of security (on a 7-point Likert scale).
  Range: 1-7 Higher score = Better outcome
Entry in nursing home | Any time within the first six months after enrolment.
  Days since enrolment when the person entered a nursing home.
  Analysed as a right censored variable. The event happening in a worse outcome. Death is treated as censoring.
(I)ADL | At enrolment and at six month follow up.
  Endpoint will be calculated as the within-subject difference in measurement between baseline and six-month follow-up for ad-hoc questions on assistance received on(I)ADL domains.
  (Instrumental) Activities of Daily Living How many of 15 activities need help to be performed? Two scores: informal caregiver help, and professional caregiver help.
  Range: 0-15 Higher value = Worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Ergo2.0, Yvoir, Belgium

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared for all collected data. Pseudonymised individual study data will undergo an anonymisation process with the help of an expert in data anonymity to ensure that no combination of data would allow re-identification of participants. The data will be publicly available on UCLouvain's public open data repository http://dataverse.uclouvain.be/.
Supporting Information: Study Protocol, ICF
Time Frame: IPD will be shared after the complete study data has been collected and anonymised (expected data: january 2026). This data will remain available on dataverse.uclouvain.be with no end date.
  ICF and study protocol will be published in a scientific journal. This data will remain available on the journal website with no end date.